CLINICAL TRIAL: NCT00091624
Title: A Phase I Study of DVd +/ CC-5013 in Relapsed Refractory Multiple Myeloma (MM)
Brief Title: A Study of Doxil, Vincristine and Decadron (DVd) +/ CC-5013 in Relapsed Refractory Multiple Myeloma (MM)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-5013-MM-011
Record Dates: First submitted 2004-09-13; First posted 2004-09-15 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Multiple Myeloma
Keywords: CC-5013; CC5013; Revlimid; Lenalidomide; Multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: CC-5013

SUMMARY:
A Phase I Study of CC-5013 in combination with Doxil, Vincristine and Decadron (DVd) in Subjects with Relapsed or Refractory Multiple Myeloma

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign an informed consent form.
* Age greater than 18 years at the time of signing the informed consent form.
* Able to adhere to the study visit schedule and other protocol requirements.
* Diagnosed with active multiple myeloma and be considered to have disease progression after at least 2 cycles of anti-myeloma treatment or have relapsed with progressive disease after treatment.
* Measurable myeloma paraprotein levels in serum (≥ 0.5g/dL) or urine (≥ 0.2 g excreted in a 24-hour collection sample).
* Eastern Cooperative Group (ECOG) Performance Status of 0-2. Performance status of 3 and 4 will be allowed if related to bony disease.
* Bilirubin < 2 x upper limits of normal (ULN).
* Liver enzymes (ALT or AST) < 3 x ULN.
* Must have adequate bone marrow function: * Absolute neutrophil count > 1,000 cells/mm3 (1.0 x 109/L) * Platelets ≥ 100,000 cells/mm3 (100 x 109/L) * Hemoglobin ≥ 8 g/dL
* Must have adequate renal function: creatinine ≤ 2.5 mg/dL.
* Must have 2-d echocardiogram indicating LVEF ≥ 50% within 42 days prior to first dose of study drug.
* Women of childbearing potential (WCBP) must have a negative serum or urine pregnancy test within 7 days of starting study drug. In addition, sexually active WCBP must agree to use adequate contraceptive methods (oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner) while on study drug. WCBP must agree to have pregnancy tests every 4 weeks while on study drug.

Exclusion Criteria:

* Severe infection requiring intravenous antibiotic treatment.
* Life expectancy of less than 3 months.
* Prior malignancy, except for adequately treated basal cell or squamous cell skin cancer, in-situ cervical cancer, or other cancer from which the subject has been disease-free for at least 5 years.
* Solitary bone or solitary extramedullary plasmacytoma as the only evidence of plasma cell dyscrasia.
* Subjects who have received > 500mg/m2 of doxorubicin alone, or Doxil® alone, or doxorubicin plus Doxil®.
* Prior treatment with CC-5013.
* Prior development of ≥ grade 2 (NCI CTC) allergic reaction/hypersensitivity while taking thalidomide.
* Prior development of a ≥ grade 3 (NCI CTC) rash or any desquamation while taking thalidomide.
* History of cardiac disease, with New York Heart Association Class II or greater.
* Uncontrolled medical problems such as diabetes mellitus, coronary artery disease, hypertension, unstable angina, arrhythmias), pulmonary, hepatic and renal diseases unless renal insufficiency is felt to be secondary to multiple myeloma.
* Any investigational agent or systemic anti-myeloma therapy within 28 days of the first dose of treatment.
* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
* Pregnant or lactating females.
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2003-03; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Knight, MD, Study Director — Celgene Corporation
Locations (1):
- Cleveland Clinic Myeloma Program, Cleveland, Ohio, United States

REFERENCES:
- [Background] Lazaryan A, Hussein MA, Reu FJ, Faiman B, Habecker B, Ann Karam M, Reed J, Hamilton K, Waksman J, Bruening K, Srkalovic G, Andresen S, Kalaycio M, Sweetenham JW, Sobecks R, Dean R, Knight R, Zeldis JB, Baz R. Mature results of MM-011: a phase I/II trial of liposomal doxorubicin, vincristine, dexamethasone, and lenalidomide combination therapy followed by lenalidomide maintenance for relapsed/refractory multiple myeloma. Am J Hematol. 2014 Apr;89(4):349-54. doi: 10.1002/ajh.23639. Epub 2014 Feb 24. PMID 24273135
- [Background] Baz R, Walker E, Karam MA, Choueiri TK, Jawde RA, Bruening K, Reed J, Faiman B, Ellis Y, Brand C, Srkalovic G, Andresen S, Knight R, Zeldis J, Hussein MA. Lenalidomide and pegylated liposomal doxorubicin-based chemotherapy for relapsed or refractory multiple myeloma: safety and efficacy. Ann Oncol. 2006 Dec;17(12):1766-71. doi: 10.1093/annonc/mdl313. Epub 2006 Sep 15. PMID 16980599